CLINICAL TRIAL: NCT07115511
Title: Combined Recanalization Therapy for Acute Large Vessel Occlusion Stroke
Acronym: CRTALVOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Gao Kaiming, DOC., Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRTALVOS2025; tianjin Huanhu hospital (Other: tianjin Huanhu hospital)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group（surgical treatment） (Experimental)
  Interventions: Procedure: Surgery
- control group（conservative therapy） (No Intervention)

INTERVENTIONS:
Procedure: Surgery — Recombined recanalization surgery
  Arms: experiment group（surgical treatment）

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of combined recanalization therapy in patients who cannot be recanalized by acute large vessel occlusive stroke. The main questions it aims to answer are:

1、Proportion of subjects with mRs score of 0-1 at 90 days after surgery

Participants will:

1、In acute large vessel occlusive stroke, if traditional means cannot be recanalized, combined recanalization surgery (including arteriotomy and thrombectomy, cerebrovascular bypass surgery) is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75.
2. According to the current guidelines, there is a MT indication.
3. Before stroke, mRS ≤2;
4. ASPECTS ≥6;
5. MCA occlusion, with or without ICA occlusion;
6. MT unsuccessful, TICI score 0-1;
7. Time from onset to craniotomy expected to be 24 hours or less;
8. Post-awakening stroke with mismatch between the infarct zone and the penumbra zone;

Exclusion Criteria:

1. Comorbid hemorrhagic vascular disease such as intracranial aneurysm or vascular malformation or other planned cerebrovascular surgery that may alter cerebral hemodynamics or lead to stroke;
2. unstable angina or myocardial infarction, congestive heart failure within the previous 6 months;
3. Pregnancy or perinatal period;
4. Hematologic disorders resulting in coagulation disorders;
5. Combination of other diseases with a life expectancy of less than 2 years; and
6. previous treatment with intracranial or extracranial vascular bypass surgery;
7. allergy to iodine or X-ray contrast media, creatinine >3.0 mg/dl or other contraindications to arteriography;
8. Uncontrolled diabetes mellitus, fasting blood sugar (FBS) >16.7 mmol/L;
9. Uncontrolled hypertension with sitting systolic blood pressure >180 mmHg or sitting diastolic blood pressure >110 mmHg;
10. Severe hepatic dysfunction, defined as serum alanine aminotransferase (ALT) and/or alanine aminotransferase (AST) >3 times the upper limit of normal;
11. Platelets <100×109 /L.
12. Received a clinical trial drug or device within 30 days prior to screening, or is participating in another clinical trial;
13. contraindication to general anesthesia or craniotomy;
14. other diseases or medical history that, in the investigator's judgment, may affect the efficacy or safety evaluation of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with mRs score of 0-1 at 90 days after surgery | 90 days after recombined recanalization surgery

SECONDARY OUTCOMES:
Changes in NIHSS score at 24 hours after surgery, 7 days after surgery, 30 days after surgery and 90 days after surgery compared with baseline; | 90 days after recombined recanalization surgery
The mRs score changed from baseline at 90 days after surgery | 90 days after recombined recanalization surgery
Change from baseline in MOCA score at 90 days after surgery | 90 days after recombined recanalization surgery
Change from baseline in MMSE score at 90 days after surgery | 90 days after recombined recanalization surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huahu Hospital, Tianjin, Tianjin Municipality, China